CLINICAL TRIAL: NCT03797716
Title: A Multi-site Randomised Controlled Trial Assessing the Effectiveness of the Little Journey App at Reducing Peri-operative Anxiety Compared to Standard Care.
Brief Title: Paediatric Peri-operative Anxiety: Does the Little Journey App Help?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 18/0197
Record Dates: First submitted 2018-11-23; First posted 2019-01-09 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Anxiety Acute; Anxiety Fear; Peri-operative; Psychological Distress; Surgery; Children, Only
Keywords: Anxiety, peri-operative, preparation, app
MeSH Terms: conditions — Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care arm (No Intervention): Participants will receive standard of care from the pre-assessment clinic until discharge.
  A typical preparatory National Health Service pathway would include: meeting a specialist nurse in the preoperative assessment clinic; a preoperative anaesthetic and surgical consultation; interaction with health play specialists on the day of surgery; and distraction interventions such as hand-held tablets during induction of anaesthesia. Participants may have inhalation or intravenous induction depending on the primary management plan of the anaesthetist in charge.
  Participants in the standard care arm will also receive a virtual reality cardboard headset, which can be taken home, personalised and decorated before use with virtual reality apps available to download from the app stores.
- Intervention arm (Experimental): Participants allocated to the intervention arm will receive the same peri-operative management as the standard care arm and will also receive an access code enabling them to use the Little Journey app in the weeks leading up to their operation. We suggest the Little Journey app is used in the days to weeks leading up to the child's operation depending on their age. On downloading the app, if parents/carers insert the age of the child and date of surgery into the Little Journey app they will be sent a push notifications reminding them when to use it according to their child's age. However, it can be used as frequently as the child and/or their parents or carers wish before the operation.
  Interventions: Device: Little Journey app

INTERVENTIONS:
Device: Little Journey app — The Little Journey app allows children to explore 360-degree hospital environments familiarising and desensitising them to areas and staff they'll see on the day of surgery. Children can "visit" the day case ward, anaesthetic and recovery rooms where their operation will occur -all while feeling safe in their own home. As the child explores the three areas, they are introduced to animated characters of staff who explain what will happen, the equipment that will be used and how they might feel. Using head tracking technology, the child triggers the animated characters by looking at them; meaning they control the pace of learning and speed at which they progress. The preparatory tool follows a pre-set story-line reflecting what happens from admission to discharge on the day of surgery.
  Arms: Intervention arm

SUMMARY:
To evaluate the clinical effectiveness of a virtual reality psychological preparation app at reducing peri-operative anxiety and its associated sequelae in children aged 3-12 years old undergoing ambulatory surgery compared to standard care.

DETAILED DESCRIPTION:
This is a phase III multi-centre randomised controlled trial evaluating the effectiveness of the Little Journey app: a pre-hospital psychological preparation tool designed for children undergoing ambulatory surgery.

Participants are pre-screened virtually through assessment of those placed on a waiting list for day case surgery at participating sites. Due to the Covid-19 pandemic, preoperative assessment clinic appointments for children undergoing ambulatory surgery have in general, moved from face-to-face appointments to telephone consultations. To enable consent and enrolment of suitable participants undergoing either telephone or face-to-face preoperative assessment, two consent pathways were developed:

Pathway 1: Remote consent. Participants are pre-screened virtually through assessment of those placed on a waiting list for day case surgery at participating sites. Pre-screening is based on the age of the child, and contingent on there being a minimum of 9 days between telephone consent and the day of planned surgery. This window has been developed to provide a minimum of 5 days of potential use time for the Little Journey app (allowing 2-3 days for the headset to arrive with the participant).

All eligible participants' parents/carers are sent a participation information sheet at least 48 hours before being approached for consent, and a copy of the consent form, by email or post. Children are also sent an information leaflet tailored to their age. A minimum of 3 working days will be provided to the parent / carer, between the research team sending them the PIS and subsequently being approached for telephone consent. Telephone consent follows a pre-approved script with opportunity provided for the parent/carer to ask questions. Families are provided with a copy of the consent form to refer to during the conversation. Telephone consent is documented on stage one of the consent form and placed in the patient notes. Written confirmation of consent (stage 2 of the consent form) is sought when the patient and carer come to hospital for surgery and before the time of transfer from the ward/outpatient are to the operating department. A copy of the signed consent form is provided to the participant's parent/carer and in the clinical notes; the original is retained in the investigator site file.

If available, at the time of consent, an assent form will be completed for children aged between 8 and 12 years of age.

Pathway 2: Face-to-face consent. Participants are pre-screened at the time of adding to a waiting list for a preoperative assessment clinic (PAC) appointment. Again, pre-screening will be based on the age of the child. All eligible participants' parents/carers are sent a PIS by email or post at least 3 working days before the planned PAC appointment. Children are also sent an information leaflet tailored to their age. Parents/carers may also be telephoned by a member of the research team informing them that the study is taking place, signposting them to the PIS, and informing them that a member of the research team will be at the PAC hoping to speak to them to offer the opportunity to take part in the trial.

At the PAC, children and their carers will undergo the standard evaluation and explanation of surgery and anaesthesia by a healthcare professional. This healthcare professional will ask if the parent/child are willing to speak with a member of the research team about the trial. If agreed, a member of the research team will then approach the parents/carers and children with a verbal explanation for the research and give them an opportunity to gain further information. If the parents/carers are content with the information provided, they will be asked to provide written consent for them and their child to be entered in the trial

Intervention Children assigned to the intervention arm will be provided with a virtual reality google cardboard headset and access code for the Little Journey app which they can use as many times as they wish before their operation. They will also receive the standard pre-operative preparation and care as per the recruiting site. In comparison, the standard care arm will receive a google cardboard virtual reality headset with suggestions of free virtual apps to use and standard pre-operative preparation and care - as defined by each participating site.

Outcome Children's anxiety will be assessed at multiple time points along the surgical journey, ranging from the preoperative assessment clinic (if occurring), ward and finally in the anaesthetic room during the induction of anaesthesia. Secondary outcome measures such as parent anxiety levels, post-hospital behavioural changes, need for rescue analgesia and antiemetics in the recovery room will be recorded.

Children's anxiety scores in those assigned to the intervention arm will undergo a further analysis assessing the impact of frequency and timing of Little Journey app use before surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 3-12 years of age on the date of parental consent to participate in the trial
2. Those undergoing surgery planned to be conducted as a day-case (surgery is defined as any therapeutic procedure taking place under the care of an anaesthetist and surgeon or dentist)
3. Requiring general anaesthetic (must be their first general anaesthetic)
4. Both child and parent able to speak / understand one of the languages available on the app
5. American Society of Anesthesiologists' physical status class I-III

   * Class I: A normal healthy patient
   * Class II: A patient with mild systemic disease
   * Class III: A patient with severe systemic disease

Note: Surgery is defined as any procedure occurring in a theatre under the care of a surgeon or dentist and an anaesthetist.

Exclusion Criteria:

1. Children aged less than 3 years of age or more than 12 years' old on the date of parental consent
2. Any child and/or parent that refuses to be part of the study
3. Patients and parents who do not speak one of the languages which are available on the app
4. Children undergoing diagnostic procedures (e.g. scans, cardiac catheterisation)
5. Any child with a visual or hearing impairments significant enough to prevent use of the intervention as decided on case-by-case basis.
6. American Society of Anesthetists physical status class IV-VI

   * Class IV: A patient with severe systemic disease that is a constant threat to life.
   * Class V: A moribund patient who is not expected to survive without the operation.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 596 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Modified Yale Pre Operative Anxiety scale - short form(m-YPAS-SF) | Day of surgery (Day 1): Measured during the induction of anaesthesia in the anaesthetic room
  An independent and blinded observer completed observational scoring tool. Children are scored in four categories: Activity, vocalisations, emotional expressivity and state of apparent arousal, according to pre-determined Likert scale observations. Each category score is divided by its highest possible score, before being added together; these scores are then divided by four and multiplied by 100, giving a value between 22.92 to 100. Higher values indicate greater anxiety levels, with scores greater than 30 typically representing clinically significant anxiety.

SECONDARY OUTCOMES:
Modified Yale Pre Operative Anxiety scale - short form(m-YPAS-SF) | Two weeks to six months before surgery: mYPAS-SF measured pre-randomisation in the Pre-Assessment clinic occurring a minimum of two-weeks before surgery, up to six-months before surgery depending on the participating research site.
  An independent and blinded observer completed observational scoring tool. Children are scored in four categories: Activity, vocalisations, emotional expressivity and state of apparent arousal, according to pre-determined Likert scale observations. Each category score is divided by its highest possible score, before being added together; these scores are then divided by four and multiplied by 100, giving a value between 22.92 to 100. Higher values indicate greater anxiety levels, with scores greater than 30 typically representing clinically significant anxiety.
  This only occurs if recruited through the Pre-Assessment clinic route.
VAS - Parent Anxiety (VAS-PA) | Two-weeks to six-months before surgery: Measured pre-randomisation in the pre-assessment clinic occurring between two-weeks to six-months before surgery date.
  A 100mm visual analogue scale assessing the current anxiety levels of parents (VAS-PA) about their child's surgery. The VAS-PA is a rapid method of assessing self-reported anxiety levels of parents before surgery. Self reported scores range from 0-100mm with higher scores signifying greater anxiety. This only occurs if recruited through the Pre-Assessment clinic route.
Modified Yale Pre Operative Anxiety scale - short form(m-YPAS-SF) | Day of Surgery (Day 1): Measured on the ward prior to surgery
  An independent and blinded observer completed observational scoring tool. Children are scored in four categories: Activity, vocalisations, emotional expressivity and state of apparent arousal, according to pre-determined Likert scale observations. Each category score is divided by its highest possible score, before being added together; these scores are then divided by four and multiplied by 100, giving a value between 22.92 to 100. Higher values indicate greater anxiety levels, with scores greater than 30 typically representing clinically significant anxiety.
VAS - Satisfaction with pre-operative information (VAS-SI) | Day of Surgery (Day 1): Measured on the ward prior to the operation on the day of surgery.
  A 100mm visual analogue scale assessing parents' satisfaction with the pre-operative information. This parent-reported score ranges from 0-100mm with higher scores signifying higher levels of satisfaction.
VAS - Compliance | Day of surgery (Day 1): Recorded immediately following observation of the induction of anaesthesia
  A 100mm visual analogue scale assessing the child's compliance during the induction of anaesthesia completed by the independent observer following observation of the induction of anaesthesia. This independent observer reported score ranges from 0-100mm with higher scores signifying higher levels of compliance.
VAS Distress | Day of surgery (Day 1): Recorded immediately following observation of the induction of anaesthesia
  A 100mm visual analogue scale assessing the child's level of distress during the induction of anaesthesia completed by the independent observer following observation of the induction of anaesthesia. This independent observer reported score ranges from 0-100mm with higher scores signifying higher levels of distress during the induction.
VAS - Parent Anxiety (VAS-PA) | Day of surgery (Day 1): Measured immediately following observation of the induction of anaesthesia.
  A 100mm visual analogue scale assessing the current anxiety levels of parents (VAS-PA) about their child's surgery. The VAS-PA is a rapid method of assessing self-reported anxiety levels of parents before surgery. Self reported scores range from 0-100mm with higher scores signifying greater anxiety.
Time to induction | Day of surgery (Day 1): Measured from entry into the anaesthetic room to entry into theatre.
  The time taken for the induction of anaesthesia (minutes)
Analgesic use | Day of surgery (Day 1): Recorded in the recovery room following surgery
  Analgesia given in the recovery room
Anti-emetic use | Day of surgery (Day 1): Recorded in the recovery room following surgery
  Anti-emetic use in the recovery room
Time to recovery | Day of surgery (Day 1): Measured from patients arrival in the recovery room until deemed ready for discharge.
  The time taken for participant to be ready for discharge back to the ward from the recovery room (minutes) as deemed by the recovery room nursing staff.
VAS- Parent satisfaction with care | Day of surgery (Day 1): Measured on the ward prior to discharge home following surgery.
  A 100mm visual analogue scale assessing parents' satisfaction with the care they received on the day of surgery. This parent-reported score ranges from 0-100mm with higher scores signifying higher levels of satisfaction.
Time to discharge | Day of surgery (Day 1): Recorded at end of day of surgery following discharge.
  The total time the participant spend in hospital from arrival on the ward to being discharged home (minutes).
Unplanned cancellations | Day of surgery (Day 1): recorded prior to attempt of induction of anaesthesia
  Incidence of unplanned cancellations on the scheduled date of surgery
Adverse events questionnaire | Day of Surgery (Day 1): Non-validated questionnaire completed immediately prior to discharge from hospital
  An assessment of the side effects of use of a virtual reality headset in both children and their parents assessed through a parent reported checkbox questionnaire.
Unplanned admissions | Day of surgery (Day 1): Recorded at end of day of surgery
  The number of participants requiring unplanned admission to hospital following surgery for any reason.
Post Hospital Behavioural Questionnaire | Day 14 post surgery: Completed at two-weeks after surgery by telephone consultation with parents/guardians
  A parent-completed eleven-point questionnaire assessing changes in their child's behaviour following surgery. Consisting of eleven items, each item is scored using a five-point Likert scale ranging from "much less than before" to " much more than before". Higher scores are suggestive of increased post hospital regressive behavioural changes.
Number of days of work/school missed | Day 14 post surgery: Completed at two-weeks after surgery by telephone consultation with parents/guardians
  The number of combined days of work missed by Parents/guardians following their child's surgery. Higher numbers are indicative of increased social costs.
Post Hospital Behavioural Questionnaire | Day 28 post surgery: Completed at four-weeks after surgery by telephone consultation with parents/guardians
  A parent-completed eleven-point questionnaire assessing changes in their child's behaviour following surgery. Consisting of eleven items, each item is scored using a five-point Likert scale ranging from "much less than before" to " much more than before". Higher scores are suggestive of increased post hospital regressive behavioural changes.
Number of days of work/school missed | Day 28 post surgery: Completed at four-weeks after surgery by telephone consultation with parents/guardians
  The number of days of school missed by children following their surgery. Higher numbers are indicative of increased social costs.

CONTACTS AND LOCATIONS:
Overall Officials: Ramani S Moonesinghe, MBBS, MRCP, FRCA, FFICM, MD, Study Chair — University College, London
Locations (17):
- United Kingdom (17):
  - Barnet Hospital, Barnet
  - Royal United Hospital Bath, Bath
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - University Hospitals Bristol and Weston NHS Trust, Bristol
  - Mid Essex Hospital (Broomfield Hospital), Chelmsford
  - Medway Maritime Hospital, Gillingham
  - Glasgow Children's Hospital, Glasgow
  - Princess Alexandra Hospital, Harlow
  - Leeds Children's hospital, Leeds
  - Royal Free Hospital, London
  - Royal London Hospital Bart's Health, London
  - University College London Hospitals, London
  - Whipps Cross Hospital Bart's Health, London
  - Royal Manchester Children's Hospital, Manchester
  - University Hospitals Plymouth, Plymouth
  - University Hospitals Southampton, Southampton
  - Torbay & South Devon, Torquay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans C, Bercades G, Ambler G, Wilson M, Brew-Graves C, Baldini C, Begum-Ali N, Williams NR, Emberton M, Fenton M, Fancourt D, Samani M, Mythen M, Moonesinghe SR. Little Journey: a phase III randomised controlled trial of a psychological preparation and education smartphone application for management of paediatric perioperative anxiety compared with standard care in children undergoing ambulatory surgery - study protocol. BMJ Open. 2025 Feb 26;15(2):e090696. doi: 10.1136/bmjopen-2024-090696. PMID 40010809